CLINICAL TRIAL: NCT06987721
Title: Comparison of the Efficacy of Radial and Focused Extracorporeal Shock-wave Therapy (ESWT) in Myofascial Pain Syndrome: Prospective, Randomized, Sham Controlled Study
Brief Title: Extracorporeal Shock-wave Therapy in Myofascial Pain Syndrome
Acronym: ESWT
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hüma Bölük Şenlikci, Associate Professor, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkent-E2-22-3033
Record Dates: First submitted 2024-09-24; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Myofacial Pain Syndrome
Keywords: Trapezius muscle; Trigger points; Pain; Therapy: pain management
MeSH Terms: conditions — Facial Neuralgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Radial ESWT: Group of participants received radial ESWT.
  Interventions: Device: Modus ESWT-Radial
- Focused ESWT: Group of participants received focused ESWT.
  Interventions: Device: Modus ESWT-Focused
- Sham group: group of participants received sham ESWT application
  Interventions: Device: Modus ESWT-Sham

INTERVENTIONS:
Device: Modus ESWT-Focused — In accordance with the literature, the ESWT adjustment is made as 1500 pulses, 0.056 mj/mm, 6 Hz for focused applications. All applications were done with the same device; Modus ESWT.
  Groups: Focused ESWT
Device: Modus ESWT-Radial — In accordance with the literature, the ESWT adjustment is made as 1500 pulses, 0.1 mj/mm, 10-16 Hz for radial applications. All applications were done with the same device; Modus ESWT.
  Groups: Radial ESWT
Device: Modus ESWT-Sham — The sham application was made in such a way that the device was set to 0 frequency and power, making only sound. All applications were done with the same device; Modus ESWT.
  Groups: Sham group

SUMMARY:
Introduction: Myofascial pain syndrome (MPS) is a syndrome characterized by painful trigger points on palpation located at certain points of common muscles of the musculoskeletal system. Active trigger points may cause spontaneous pain and many other consequences that affect quality of life and loss of work force. Extracorporeal shock-wave therapy (ESWT) is a treatment method performed with the help of acoustic waves created outside the body and used in musculoskeletal problems. There are radial or focused waves that are commonly used in ESWT. In Focused ESWT (F-ESWT), the depth of the body part to be injured can be adjusted. Thus, penetration into the tissue is better than radial waves. Radial ESWT (R-ESWT), on the other hand, has a more superficial effect, and its spread in liquids with a density similar to tissues is half that of focused ESWT. It has been shown in previous studies that radial and focused ESWT waves applied to trigger points in the upper trapezius fibers reduce reflected and local pain in myofascial pain syndrome. The aim of this study is to compare the effectiveness of radial and focused ESWT types on trigger points in trapezoidal upper fibers in myofascial pain syndrome.

Methods: This prospective,sham-controlled double-blind study was carried out with total of 57 patients. They were randomized into 3 groups and received R-ESWT, F-ESWT and sham protocols for 10 sessions. Patients were evaluated and compared with Numerical rating scale (NRS), Health assessment Questionnaire (HAQ) and Beck Depression Scale (BDI) before treatment, just post treatment, 1st month, 3nd month and 6th month after treatment completed.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a syndrome characterized by painful trigger points on palpation located at certain points of common muscles of the musculoskeletal system. Pain on palpation tends to radiate and is sometimes even accompanied by sensory symptoms (such as paresthesia) or autonomic findings (piloerection, sweating, etc.). Trigger points can be either latent or active. Active trigger points may cause spontaneous pain, while latent trigger points are more commonly manifested as pain radiating with palpation. Latent trigger points tend to turn into active trigger points as a result of acute stresses, microtraumas or postural disorders, and the trapezius muscle is the most common muscle in which myofascial trigger points are seen. Myofascial pain syndrome can cause many consequences such as disturbances in daily living acitivities, decrease in quality of life and loss of work force. It can also accompany anxiety and depression . Pharmacological therapy can be used in the treatment, since stretching exercises, dry needling, acupuncture or physical therapy modalities are another effective treatment options for patients who are not willing to use drugs or have co-morbidities .

Extracorporeal shock-wave therapy (ESWT) is a kind of physical therapy method performed with the help of acoustic waves created outside the body. It is frequently used in musculoskeletal conditions. Its effectiveness has been demonstrated in disorders such as calcaneal spur, lateral epicondylitis, calcific tendinitis, myofascial pain syndrome, and fibromyalgia .

Radial or focused waves are commonly used in application of ESWT. In Focused ESWT (F-ESWT), the depth of the body part to be injured can be adjusted. Thus, penetration into the tissue is better than radial waves. Radial ESWT (R-ESWT), on the other hand, has a more superficial effect, and its spread in liquids with a density similar to tissues is half that of F-ESWT . However some side effects were identified during the ESWT procedure, both wave types are thought to be safe and widely used.

It has been shown in previous studies that radial and focused ESWT waves applied to trigger points in the upper trapezius fibers reduce reflected and local pain in myofascial pain syndrome. The effectiveness of these waves has been evaluated in studies many times but the effectiveness of the two wave types has not been compared in patients with trigger points in the trapezius upper fibers in myofascial pain syndrome. The aim of this study is to compare the efficacy of R-ESWT and F-ESWT types on trigger points in trapezoidal upper fibers in myofascial pain syndrome.

This prospective, sham-controlled and double-blind study was carried out at Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital. Fifty nine male and/or female patients enrolled the study initially. The study protocol is compatible with Helsinki declaration and approved by Ankara Bilkent City Hospital Ethics Committee (Approval number: E2-22-3033). Written and oral informed consents were obtained from the participants before allocation.

Participants were diagnosed as MPS according to Travell and Simons' 5 major and 3 minor criteria. Major criteria were 1) localized spontaneous pain 2) presence of spontaneous pain and/or changed sensation in referred pain area 3) palpable bands in muscle 4) sharp tenderness along the taut bands 5) measurable limitation in range of motion. Minor criteria were 1) pain or change in sensation caused by touching the taut bands 2) Presence of a local twitch response in the muscle upon needle insertion 3) reduced pain after stretching or injection of taut bands. Five major and at least 1 minor criteria are needed for MPS diagnosis .

Inclusion criteria were 1) Patients aged between 18-70 years with myofascial pain syndrome and active trigger points in the trapezius upper fibers 2) Pain related to trapezius muscle trigger points were > 4 according to numerical rating scale (NRS).

Exclusion criteria were 1) revealed any cervical disc herniation (protrusion or extrusion) that cause cervical root compression showed with magnetic resonance imaging and/or radicular pain with motor or sensory deficit 2) Presence of neurological and rheumatological disorders and/or malignancy 3) Detected cognitive impairment according to mini mental test (mini mental test score <23) 4) Acute systemic infection or any other diseases that effect general condition 5) participants have any open wound or sensory deficit in the application area.

Patients who met inclusion criteria were included in the study. Randomization was done with a software system and totally 59 patients were enrolled (20 R-ESWT, 19 F-ESWT, 20 sham). One patient did not come to follow-ups and one patient left the study before the completion of sessions and eventually 57 patients were completed the study (Figure 1). Sociodemographic and clinical characteristics of the patients were recorded before the procedure.

Exercise program for strecthing exercises of trapezius muscle were given for all the participants for 4 weeks. Weekly remindings were done with telephone calls and face-to-face follow-ups. All ESWT applications were made in a total of 4 sessions with one week between them by one of the researcher physician. Patients included in the study were evaluated at the beginning of the study (pre-treatment), just after completion of ESWT sessions, at 1st month, 3rd month and 6th month after the end of 4 sessions in terms of pain, functionality and depression.

In accordance with the literature, the ESWT adjustment is made as 1500 pulses, 0.1 mj/mm, 10-16 Hz for radial applications, and 1500 pulses, 0.056 mj/mm, 6 Hz for focused applications. The sham application was made in such a way that the device was set to 0 frequency and power, making only sound. All applications were done with the same device; Modus ESWT.

Randomization and blinding Patients diagnosis were done by the same physician. Informed consent were obtained and patients were informed that they were not going to be able to aware of the group they participate due to the type of the study, in addition first evaluations were done with a face to face interview by the same physician.

After diagnosed as MPS, patients were randomized by a data entry staff with a software. Another physician who had done all ESWT applications were informed about the application type by the staff according to that software. After all sessions were completed, first evaluator physician who is blind to application type, assessed patients at follow-ups.

Numerical Rating Scale (NRS) Numerical rating scale (NRS) is used by patients to perform a self-assessment of pain intensity associated with myofascial pain syndrome. Higher scores indicates more pain related to trigger points of upper trapezius muscle fibers .

Beck Depression Inventory (BDI) Beck Depression Inventory (BDI) is used to evaluate the characteristics of depression and anxiety. BDI consists of 21 questions, higher scores imply increased depression symptom severity .

Health Assesment Questionnaire (HAQ) This questionnaire has 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each item is between 0-3 (0=without any difficulty, 3=unable to do). Higher scores indicate worse health condition according to the patient's own reports.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18-70 years with myofascial pain syndrome and active trigger points in the trapezius upper fibers
2. Pain related to trapezius muscle trigger points were > 4 according to numerical rating scale (NRS)

Exclusion Criteria:

1. Revealed any cervical disc herniation (protrusion or extrusion) that cause cervical root compression showed with magnetic resonance imaging and/or radicular pain with motor or sensory deficit
2. Presence of neurological and rheumatological disorders and/or malignancy 3. Detected cognitive impairment according to mini mental test (mini mental test score <23)

4. Acute systemic infection or any other diseases that effect general condition 5. Participants have any open wound or sensory deficit in the application area.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18-75 years old with myofascial pain syndrome and that have trigger points in upper trapezius muscles were participated in the study
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | Before treatment, just post treatment, 1st month, 3nd month and 6th month after treatment completed.
  Numerical rating scale (NRS) (0-10 scores) is used by patients to perform a self-assessment of pain intensity associated with myofascial pain syndrome. Higher scores indicates more pain related to trigger points of upper trapezius muscle fibers

SECONDARY OUTCOMES:
Beck Depression Inventory | Before treatment, just post treatment, 1st month, 3nd month and 6th month after treatment completed.
  Beck Depression Inventory (BDI) is used to evaluate the characteristics of depression and anxiety. BDI consists of 21 questions, higher scores imply increased depression symptom severity. Scores are between 0-63 points.
Health Assessment Questionnaire | Before treatment, just post treatment, 1st month, 3nd month and 6th month after treatment completed.
  This questionnaire has 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each item is between 0-3 (0=without any difficulty, 3=unable to do). Higher scores indicate worse health condition according to the patient's own reports

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD is going to be shared in submission process
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD is going to be shared in submission process
Access Criteria: other researchers

REFERENCES:
- [Background] Schmitz C, Csaszar NB, Milz S, Schieker M, Maffulli N, Rompe JD, Furia JP. Efficacy and safety of extracorporeal shock wave therapy for orthopedic conditions: a systematic review on studies listed in the PEDro database. Br Med Bull. 2015;116(1):115-38. doi: 10.1093/bmb/ldv047. Epub 2015 Nov 18. PMID 26585999
- [Background] Paoletta M, Moretti A, Liguori S, Toro G, Gimigliano F, Iolascon G. Efficacy and Effectiveness of Extracorporeal Shockwave Therapy in Patients with Myofascial Pain or Fibromyalgia: A Scoping Review. Medicina (Kaunas). 2022 Jul 28;58(8):1014. doi: 10.3390/medicina58081014. PMID 36013480
- [Background] Urits I, Charipova K, Gress K, Schaaf AL, Gupta S, Kiernan HC, Choi PE, Jung JW, Cornett E, Kaye AD, Viswanath O. Treatment and management of myofascial pain syndrome. Best Pract Res Clin Anaesthesiol. 2020 Sep;34(3):427-448. doi: 10.1016/j.bpa.2020.08.003. Epub 2020 Aug 8. PMID 33004157
- [Background] Tasoglu O, Sahin Onat S, Boluk H, Tasoglu I, Ozgirgin N. Comparision of two different dry-needling techniques in the treatment of myofascial pain syndrome. Agri. 2017 Jan;29(1):9-16. doi: 10.5505/agri.2016.38991. PMID 28467572
- See also: Study Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4674007/pdf/ldv047.pdf